CLINICAL TRIAL: NCT05528120
Title: Food Effect Study on the Pharmacokinetics of VC004 Capsules in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VC004-103
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Locally Advanced or Metastatic Solid Tumor Harboring an NTRK Gene Fusion
Keywords: healthy subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KG (Experimental)
  Interventions: Drug: VC004 Capsules
- GK (Experimental)
  Interventions: Drug: VC004 Capsules

INTERVENTIONS:
Drug: VC004 Capsules — Oral administration after fasting/high-fat meal
  Arms: KG
Drug: VC004 Capsules — Oral administration after high-fat/fasting meal
  Arms: GK

SUMMARY:
This study will adopt a randomized, open-label, two-period, 2-way crossover design to evaluate pharmacokinetics of a single oral dose of VC004 capsules under fasting and fed conditions in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent before study, and fully understand the study content, process and possible adverse reactions;
2. Able to complete the study in compliance with the protocol;
3. Subject (including partner) is willing to voluntarily take effective contraceptive measures from screening through 6 months after the last dose of study drug (see Appendix 5 for details);
4. Male and female subjects between the ages of 18 and 45 years, inclusive;
5. At least 50.0kg for male subjects, 45.0kg for female subjects, with a Body Mass Index (BMI= Weight/Height2) between 19.0-26.0 kg/m2, inclusive;

Exclusion Criteria:

1. More than 5 cigarettes per day on average within 3 months prior to screening;
2. History of sensitivity to drugs similar to the study drug;allergic constitution (e.g. allergy to two or more kinds of drugs and food );
3. History of drug and/or alcohol abuse (alcoholism defined as: drinking 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine); history of drug abuse or or have used drugs within the past five years;
4. Donation or loss of a significant volume of blood (> 450 mL) within 3 months prior to screening;
5. History of difficulties in swallowing or any history of gastrointestinal, liver, kidney disease (whether cured or not) or surgery that affects drug absorption or excretion within 6 months prior to screening;
6. Those who Have taken strong inhibitors and / or inducers of liver metabolic enzymes (CYP1A2, 2A6, 2b6, 2c8, 2c19, 3A4 and 3A5) within 28 days before the first administration :strong inhibitors of liver metabolic enzymes such as ciprofloxacin, clopidogrel, itraconazole, ketoconazole, ritonavir, oleandomycin etc., strong inducers of liver metabolic enzymes such as rifampicin, carbamazepine, phenytoin sodium, St. John's wort, etc; Those who Have taken inhibitors and inducers of P-gp, MRPs, BCRP, OATP and other transporters and transporters within 28 days before the first administration; See Appendix 6 for details;
7. Intake of any prescription drugs, over-the-counter drugs, vitamin or herbal medicine within 14 days prior to receiving study drug;
8. Taking foods that affect CYP3A4 metabolism, such as grapefruit or drinks containing grapefruit within 2 weeks before the first drug administration, or taking high-intensity physical exercises (such as strength training, aerobic training and football playing) within 7 days before the first drug administration, or any other factors that affect drug absorption, distribution, metabolism and excretion;
9. Recent major changes in diet or exercise habits within 7 days before the first medication;
10. Participated in other clinical trials within 3 months before screening (if the subject withdraws from the study before treatment, i.e. has not been randomized or received treatment, he or she can be enrolled in the study);
11. Those who cannot tolerate high-fat meals or have special requirements for diet and cannot accept unified diet；
12. A clinically significant vital signs abnormality during screening (body temperature (axillary temperature) < 36.0 ℃ or > 37.0 ℃; Pulse < 60bpm or > 100bpm; Systolic blood pressure <90mmhg or ≥ 140mmHg, diastolic blood pressure <60mmhg or ≥ 90mmHg);
13. A clinically significant 12-lead ECG abnormality;
14. Positive test results of blood pregnancy or is lactating for female subjects;
15. Any clinically significant abnormalities/findings in laboratory tests, or any clinically significant disease including but not limited to gastrointestinal, renal, hepatic, neurological system, blood, endocrine, tumor, lung, immune, mental, or cardiovascular and cerebrovascular diseases;
16. Positive test results for viral hepatitis (including hepatitis B and C), HIV antibody or syphilis antibody during screening;
17. Acute illness or concomitant medication from screening to the first dosing of study medication;
18. Consumption of chocolate or any food or beverages containing caffeine or (rich containing) xanthine within 24 h prior to receiving the first dosing of study medication;
19. Consumption of any product containing alcohol within 24 h prior to receiving the first dosing of study medication, or positive results from a screen for alcohol;
20. Positive results from a screen for urine drug test;
21. Cannot tolerate venipuncture and have a history of needle and blood sickness;
22. Subjects were vaccinated within 4 weeks prior to screening, or planned to be vaccinated during the trial;
23. Any condition which in the opinion of Investigator is not suitable for subjects to participate in the study or who are not suitable to participate according to the epidemic prevention and control requirements of the research center.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day1-Day8
Peak time(Tmax) | Day1-Day8
Area Under the Curve From Time Zero to Last Quantifiable Concentration(AUC） | Day1-Day8

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital,Affiliated to Southeast University, Nanjing, Jiangsu, China